CLINICAL TRIAL: NCT04400799
Title: Enoxaparin for Primary Thromboprophylaxis in Ambulatory Patients With Coronavirus: The Multicenter Randomized Controlled Ovid Trial
Brief Title: Enoxaparin for Primary Thromboprophylaxis in Ambulatory Patients With COVID-19
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: due to results from interim analysis
Sponsor: University of Zurich (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other); Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Basel, Switzerland (Other); Oncology Institute of Southern Switzerland (Other); Clinica Luganese Moncucco (Other); University Hospital Freiburg (Other); Mainz University (Other)
Responsible Party: Principal Investigator, Nils Kucher, Prof. Dr. med., University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVID Trial
Record Dates: First submitted 2020-05-15; First posted 2020-05-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: COVID-19; Pulmonary Embolism, Deep Vein Thrombosis
MeSH Terms: conditions — COVID-19; Pulmonary Embolism; Venous Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Enoxaparin (Clexane®) will be given at the recommended dose of 4,000 IU antiXa activity (40 mg/0.4 ml) once daily by SC injection for 14 days.
  Interventions: Drug: Enoxaparin 40Mg/0.4Ml Inj Syringe 0.4Ml
- Control Group (No Intervention): No study drug

INTERVENTIONS:
Drug: Enoxaparin 40Mg/0.4Ml Inj Syringe 0.4Ml — daily incetion s.c. for 14 days
  Arms: Test Group

SUMMARY:
The OVID study will show whether prophylactic-dose enoxaparin improves survival and reduces unplanned hospitalizations in ambulatory patients aged 50 or older diagnosed with COVID-19, a novel viral disease characterized by severe systemic, pulmonary, and vessel inflammation and coagulation activation.

DETAILED DESCRIPTION:
The following points represent, in summary, the rationale for studying the use of thromboprophylaxis in ambulatory patients with COVID-19:

1. The risk of thromboembolic events in patients with COVID-19 during anticoagulant prophylaxis exceeds that observed in medical patients, usually <3%, even in the presence of seasonal viral infections
2. The cumulative risk of VTE in hospitalized COVID-19 patients is at least 20%, but possibly higher, as described in several publications
3. The absolute VTE risk in COVID-19 patients requiring intensive care is 69% if screening strategies are implemented
4. Half of the VTE events, mostly PE, were diagnosed at hospital admission, suggesting that these events developed during the quarantine period.

Our hypothesis is that early thromboprophylaxis may prevent or limit coagulopathy, and reduce thromboembolic complications leading to hospitalization or death, in the presence of a mild COVID disease among outpatients.

The study will be conducted as a multicentre randomized open-label controlled trial. In the study, a total of 1,000 adult patients aged 50 or older with COVID-19 and candidates to ambulatory treatment will be randomized to receive enoxaparin 40 mg sc qD or no treatment for a total of 14 days. The primary outcome will be assessed within 30 days of enrolment.

We implemented two logistical solutions to integrate the process of SARS-CoV2 testing, pre-screening, screening (hot-line and flyers), in-hospital recruitment, enrolment and randomization/allocation. A nationwide OVID Hot-Line telephone number will be made available in 3 languages (German, French, Italian) for interested patients or test centers to contact the Hot-Line. Standard hygiene precautions will be met at the study centers to avoid spreading of SARS-CoV2 among other patients or health care workers. Principles of patient and investigator safety will be applied. Standard procedures concerning privacy, discussion with patients on details of the study, collection of informed consent, and instruction on how to administer the study medication will be maintained in conformity with GCP recommendations. This will also include outcome measurements to be conducted by telephone with standardized questionnaire.

Enoxaparin (Clexane®) will be given at the recommended dose of 4,000 IU antiXa activity (40 mg/0.4 ml) once daily by SC injection for 14 days.

A single interim analysis is planned at time when the outcomes of 50% of the patients (n=460 plus drop-outs) have been observed (anticipated in February 2022).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50 years or older with a positive test for SARS-CoV2 in the past 5 days and eligible for ambulatory treatment.
2. Presence of respiratory symptoms (i.e. cough, sore throat, or shortness of breath) or body temperature >37.5° C.
3. Ability of the patient to travel to the study center by private transportation, performed either by accompanying person from same household or by the patient him/herself
4. Ability to comply with standard hygiene requirements at the time of in-hospital visit, including a face mask and hand disinfectant.
5. Ability to walk from car to study center or reach it using a wheel chair transport with the help of an accompanying person from the same household also complying with standard hygiene requirements.
6. Ability to self-administer prefilled enoxaparin injections after instructions received at the study center or availability of a person living with the patient to administer enoxaparin.

Exclusion Criteria:

1. Any acute or chronic condition posing an indication for anticoagulant treatment, e.g. atrial fibrillation, prior VTE, acute confirmed symptomatic VTE, acute coronary syndrome.
2. Anticoagulant thromboprophylaxis deemed necessary in view of the patient's history, comorbidity or predisposing strong risk factors for thrombosis:

   1. Any of the following events occurring in the prior 30 days: fracture of lower limb, hospitalization for heart failure, hip/knee replacement, major trauma, spinal cord injury, stroke,
   2. previous VTE,
   3. histologically confirmed malignancy, which was diagnosed or treated (surgery, chemotherapy, radiotherapy) in the past 6 months, or recurrent, or metastatic, or inoperable.
3. Any clinically relevant bleeding (defined as bleeding requiring hospitalization, transfusion, surgical intervention, invasive procedures, occurring in a critical anatomical site, or causing disability) within 30 days prior to randomization or sign of acute bleeding.
4. Intracerebral bleeding at any time in the past or signs/symptoms consistent with acute intracranial hemorrhage.
5. Hemoglobin <8 g/dL and platelet count <50 x 109 cells/L confirmed by recent laboratory test (<90 days).
6. Subjects with any known coagulopathy or bleeding diathesis, including known significant liver disease associated with coagulopathy.
7. Severe renal insufficiency (baseline creatinine clearance <30 mL/min calculated using the Cockcroft-Gault formula) confirmed by recent laboratory test (<90 days).
8. Contraindications to enoxaparin therapy, including prior heparin-induced thrombocytopenia and known hypersensitivity.
9. Current use of dual antiplatelet therapy.
10. Participation in other interventional studies over the past 30 days.
11. Non-compliance or inability to adhere to treatment or lack of a family environment or support system for home treatment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-04-12 (Actual)

PRIMARY OUTCOMES:
hospitalizations | 30 days
all-cause death | 30 days

SECONDARY OUTCOMES:
Number of cardiovascular events | within 14 days, 30 days, and 90 days of randomization
  including deep vein thrombosis (including catheter-associated), pulmonary embolism, myocardial infarction/myocarditis, arterial ischemia including mesenteric and extremities, acute splanchnic vein thrombosis, or ischemic stroke
any hospitalizations | within 14 days, 30 days, and 90 days of randomization
all-cause death | within 14 days, 30 days, and 90 days of randomization
Net clinical benefit | within 14 days, 30 days, and 90 days of enrolment.
  measured by number of cardiovascular events, and major bleeding
Disseminated intravascular coagulation | within 14 days, 30 days, and 90 days of enrolment
  ISTH criteria, in-hospital diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof., Principal Investigator — University of Zurich
Locations (8):
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Johannes Gutenberg-Universität Mainz, Mainz
- Switzerland (6):
  - University Hospital Basel, Basel
  - Clinic of Hematology, Oncology Institute of Southern Switzerland, Bellinzona
  - University Hospital Bern, Bern
  - Hôpitaux Universitaires Genève, Geneva
  - Clinica Luganese Moncucco, Lugano
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523
- [Derived] Barco S, Voci D, Held U, Sebastian T, Bingisser R, Colucci G, Duerschmied D, Frenk A, Gerber B, Gotschi A, Konstantinides SV, Mach F, Robert-Ebadi H, Rosemann T, Simon NR, Spechbach H, Spirk D, Stortecky S, Vaisnora L, Righini M, Kucher N; OVID investigators. Enoxaparin for primary thromboprophylaxis in symptomatic outpatients with COVID-19 (OVID): a randomised, open-label, parallel-group, multicentre, phase 3 trial. Lancet Haematol. 2022 Aug;9(8):e585-e593. doi: 10.1016/S2352-3026(22)00175-2. Epub 2022 Jun 30. PMID 35779558
- [Derived] Barco S, Bingisser R, Colucci G, Frenk A, Gerber B, Held U, Mach F, Mazzolai L, Righini M, Rosemann T, Sebastian T, Spescha R, Stortecky S, Windecker S, Kucher N. Enoxaparin for primary thromboprophylaxis in ambulatory patients with coronavirus disease-2019 (the OVID study): a structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Sep 9;21(1):770. doi: 10.1186/s13063-020-04678-4. PMID 32907635